CLINICAL TRIAL: NCT06078930
Title: A Multi-center Observational Clinical Study on the Development of Artificial Intelligence-Based Gastric Cancer Screening and Diagnosis Technology Using Multi-Omics Analysis of Tongue Imaging and Tongue Coating
Brief Title: Development of Novel Gastric Cancer Screening and Diagnosis Technologies Using Tongue Imaging and Study of Tongue Image Changes Mechanisms
Status: Recruiting | Type: Observational
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: Sichuan Cancer Hospital and Research Institute (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Wenzhou Medical University (Other); Fujian Cancer Hospital (Other Government); RenJi Hospital (Other); Tongde Hospital of Zhejiang (Unknown); Kecheng District People's Hospital (Unknown); Yueyang Central Hospital (Other); Shandong Cancer Hospital and Institute (Other); Shanxi Province Cancer Hospital (Other); Liaoning Cancer Hospital & Institute (Other); Harbin Cancer Hospital (Unknown); Yuhang District People's Hospital (Unknown); Hainan Cancer Hospital (Other); Zigong Fourth People's Hospital (Unknown); Henan University of Science and Technology (Other); Shangyu People's Hospital of Shaoxing City (Unknown); Red Cross Hospital, Hangzhou, China (Other); The Affiliated Hospital of Hangzhou Normal University (Other); Xiaoshan District First People's Hospital (Unknown); Xianju County People's Hospital (Unknown); Lin'an District First People's Hospital (Unknown); First Affiliated Hospital of Wenzhou Medical University (Other); Wenzhou Central Hospital (Other); The Third Affiliated Hospital of Wenzhou Medical University (Other); Leqing City People's Hospital (Unknown); The Affiliated Hospital of Medical School of Ningbo University (Unknown); Cixi City People's Hospital (Unknown); Mingzhou Hospital, Zhejiang University (Unknown); Fourth Hospital of Ningbo City (Unknown); Fenghua District People's Hospital (Unknown); Fenghua Traditional Chinese Medicine Hospital, Ningbo City (Unknown); Xikou Hospital, Fenghua District, Ningbo City (Unknown); Chengdu University of Traditional Chinese Medicine (Other); Guang'an Hospital, Affiliated to Chengdu University of Traditional Chinese Medicine (Unknown); Jiangsu Cancer Institute & Hospital (Other); Jiangsu Provincial People's Hospital (Other); The First People's Hospital of Changzhou (Other); The First Affiliated Hospital of Soochow University (Other); Jiangsu Provincial Hospital of Traditional Chinese Medicine (Unknown); Zidong Campus of Jiangsu Provincial Hospital of TCM (Unknown); Wuxi Traditional Chinese Medicine Hospital (Unknown); First Affiliated Hospital of Harbin Medical University (Other); The First Affiliated Hospital of Anhui Medical University (Other); Peking University Cancer Hospital & Institute (Other); Xijing Hospital (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Xiangya Hospital of Central South University (Other); Yunnan Cancer Hospital (Other); Chongqing University Cancer Hospital (Other); Gansu Cancer Hospital (Other); Fudan University (Other); Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); First Affiliated Hospital of Guangxi Medical University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Huzhou Central Hospital (Other); Zhoushan Hospital, Zhejiang (Unknown)
Responsible Party: Principal Investigator, Xiangdong Cheng, MD, Zhejiang Cancer Hospital
Other Study IDs: IRB-2021-289
Record Dates: First submitted 2023-10-05; First posted 2023-10-12 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Gastric Cancer; Tongue Images; Diagnosis
MeSH Terms: conditions — Stomach Neoplasms; Disease | interventions — Defecation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with gastric cancer
  Interventions: Diagnostic Test: Tongue imaging, tougue coating, saliva, gastric juice, and feces
- Healthy participants
  Interventions: Diagnostic Test: Tongue imaging, tougue coating, saliva, gastric juice, and feces

INTERVENTIONS:
Diagnostic Test: Tongue imaging, tougue coating, saliva, gastric juice, and feces — Tongue images, coating, saliva, gastric juice, and feces on the tongue and clinical data of patients with gastric cancer and healthy participants will be collected.

SUMMARY:
In this study, the investigators will prospectively recruit 100,000 individuals, including gastric cancer patients who have not undergone any anti-tumor treatment and non-gastric cancer participants. The investigators will construct a diagnostic model for malignant tumors based on the combination of tongue imaging, tongue coating, saliva, gastric juice, and fecal multi-omics data (including metagenomics, proteomics, metabolomics, etc.). Additionally, the study will explore the relationship between oral, gastric, and intestinal microbiota and the development of malignant tumors.

DETAILED DESCRIPTION:
Patients with gastric cancer were recruited through outpatient clinics, endoscopy units, and inpatient departments of various centers, with all patients requiring a histopathological diagnosis. Non-gastric cancer participants were sourced from community health check-ups, outpatient clinics, and endoscopy units affiliated with these centers.

ELIGIBILITY:
Inclusion Criteria for Gastric Cancer Patients:

* 18≤age≤90
* Histologically or cytologically confirmed gastric cancer
* No prior chemotherapy, radiotherapy, biotherapy, immunotherapy or other anti-tumor treatment for gastric cancer
* Subject volunteers to join the study, Signs informed consent, has good compliance and can cooperate with follow-up

Exclusion Criteria for Gastric Cancer Patients:

* Two or more kinds of malignant tumors at the same time
* Gastric cancer that has been treated by chemotherapy, radiotherapy, biotherapy, immunotherapy or other anti-tumor therapy
* The use of glucocorticoids and antibiotics in the past three months
* History of long-term medication
* Presence of oral diseases such as tooth and gum diseases
* Subjects who had other factors that might force them to terminate the research ahead of time, such as the development of other severe disease (including mental disease) that required combined treatment, seriously abnormal laboratory examination value, and family or social factors that might affect the subject safety or experimental data collection, as judged by the researchers

Inclusion Criteria for Healthy Participants:

* 18≤age≤90
* Willingness to participate in the study, signing an informed consent form, and demonstrating good compliance

Exclusion Criteria for Healthy Participants:

* History of malignant tumors
* The use of glucocorticoids and antibiotics in the past three months
* History of long-term medication
* Presence of oral diseases such as tooth and gum diseases
* Subjects who had other factors that might force them to terminate the research ahead of time, such as the development of other severe disease (including mental disease) that required combined treatment, seriously abnormal laboratory examination value, and family or social factors that might affect the subject safety or experimental data collection, as judged by the researchers

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Histologically or cytologically confirmed gastric cancer, and no prior chemotherapy, radiotherapy, biotherapy, immunotherapy or other anti-tumor treatment for malignant tumor. Gastric cancer patients and healthy participants should not have the following conditions: the use of glucocorticoids and antibiotics in the past three months, a history of long-term medication, as well as oral diseases such as tooth and gum diseases.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The differences in tongue images, tongue coating, saliva, gastric juice, and fecal samples between patients with gastric cancer and healthy individuals will be systematically analyzed. | 5 years
The differences of the clinical information between patients with gastric cancer and healthy participants. | 5 years
  These data of gastric cancer group included age, sex, height, weight, family history, smoking, drinking, TNM staging, tumor location, tumor size, pathological type, grade of differentiation, expression of Her2, nerve invasion, vascular tumor thrombus, lauren type and and blood tumour markers, and these data of healthy participants group included age, sex, height, weight, smoking, drinking and blood tumour markers.
Overall Survival (OS) | 5 years

SECONDARY OUTCOMES:
Disease Free Survival (DFS) | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
We currently have no plans to share individual participant data (IPD) with other researchers.

REFERENCES:
- [Background] Yuan L, Yang L, Zhang S, Xu Z, Qin J, Shi Y, Yu P, Wang Y, Bao Z, Xia Y, Sun J, He W, Chen T, Chen X, Hu C, Zhang Y, Dong C, Zhao P, Wang Y, Jiang N, Lv B, Xue Y, Jiao B, Gao H, Chai K, Li J, Wang H, Wang X, Guan X, Liu X, Zhao G, Zheng Z, Yan J, Yu H, Chen L, Ye Z, You H, Bao Y, Cheng X, Zhao P, Wang L, Zeng W, Tian Y, Chen M, You Y, Yuan G, Ruan H, Gao X, Xu J, Xu H, Du L, Zhang S, Fu H, Cheng X. Development of a tongue image-based machine learning tool for the diagnosis of gastric cancer: a prospective multicentre clinical cohort study. EClinicalMedicine. 2023 Feb 6;57:101834. doi: 10.1016/j.eclinm.2023.101834. eCollection 2023 Mar. PMID 36825238
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Wang FH, Zhang XT, Li YF, Tang L, Qu XJ, Ying JE, Zhang J, Sun LY, Lin RB, Qiu H, Wang C, Qiu MZ, Cai MY, Wu Q, Liu H, Guan WL, Zhou AP, Zhang YJ, Liu TS, Bi F, Yuan XL, Rao SX, Xin Y, Sheng WQ, Xu HM, Li GX, Ji JF, Zhou ZW, Liang H, Zhang YQ, Jin J, Shen L, Li J, Xu RH. The Chinese Society of Clinical Oncology (CSCO): Clinical guidelines for the diagnosis and treatment of gastric cancer, 2021. Cancer Commun (Lond). 2021 Aug;41(8):747-795. doi: 10.1002/cac2.12193. Epub 2021 Jul 1. PMID 34197702
- [Background] Li MY, Zhu DJ, Xu W, Lin YJ, Yung KL, Ip AWH. Application of U-Net with Global Convolution Network Module in Computer-Aided Tongue Diagnosis. J Healthc Eng. 2021 Nov 18;2021:5853128. doi: 10.1155/2021/5853128. eCollection 2021. PMID 34840700